CLINICAL TRIAL: NCT03577561
Title: Technology Enhanced Learning and Proficiency Based Progression to Investigate and Mitigate Blood Sampling Errors Including 'Wrong Blood in Tube' in Our Hospitals; Can we Improve Patient Safety and Reduce Resource Wastage?
Brief Title: Proficiency Based Training to Investigate Blood Sampling Errors Including WBIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patrick Henn (Other)
Collaborators: Cork University Hospital (Other)
Responsible Party: Sponsor-Investigator, Patrick Henn, Investigator, University College Cork
Organization: University College Cork (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 1820
Record Dates: First submitted 2018-04-30; First posted 2018-07-05 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Blood Transfusion Complication; Wrong Blood in Tube; Pre Analytical Blood Sample Errors
MeSH Terms: conditions — Transfusion Reaction | interventions — Phlebotomy

STUDY DESIGN:
Intervention Model Description: Control group A: 1 -year historical data (2016/2017) The blood sampling error rate in the interns receiving PBP training in 2018 will be compared to historical data on doctors who would have received whatever training they would normally undergo as a part of their existing training program. It will not differ from what they would normally receive at that institution.
  Control group B (2017/2018) In a pilot project in July 2017, 46 interns received the phlebotomy PBP training at CUH. The error rates in the interns in 2017 will be compared to the newly trained interns in 2018 to determine the effectiveness of the training over time.
  Interventional Group:
  The blood sampling error rate in those doctors in training given the improved proficiency based progression training under investigation from March 30th 2018
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group A (No Intervention): Control group A: 1 -year historical data (2016/2017) The blood sampling error rate in the interns receiving proficiency based progression training in 2018 will be compared to historical data on doctors who would have received whatever training they would normally undergo as a part of their existing training program. It will not differ from what they would normally receive at that institution.
- Control Group B (Active Comparator): Control group B (2017/2018) In a pilot project in July 2017, 46 interns received the phlebotomy proficiency based progression training at CUH. The error rates in the interns in 2017 will be compared to the newly trained interns in 2018 to determine the effectiveness of the training over time. The intervention is the proficiency based progression training programme in phlebotomy.
  Interventions: Other: Proficiency Based Progression Training in Phlebotomy
- Interventional Group (Active Comparator): The blood sampling error rate of doctors in training provided with the intervention i.e. improved proficiency based progression training programme will be analysed from July 10th 2018 until the study ends.
  The proficiency based progression training will consist of an online eLearning module to teach the doctors the correct process to take blood in the hospital. The doctors will then have to attend a face to face training day on a simulation ward where they will be asked to take blood according to a metric of 77 steps with less than 13 errors and no critical errors. Finally, the doctors will be observed taking blood on the ward and again must take it to a proficient standard.
  Interventions: Other: Proficiency Based Progression Training in Phlebotomy

INTERVENTIONS:
Other: Proficiency Based Progression Training in Phlebotomy — Trainees will receive an online didactic education package and a simulation skill training module. Both of these education and training platforms will be derived from the procedure characterisation and benchmarked on experienced practitioner's performance. Trainees will be required to engage with the education and training platforms in a process of deliberate practice learning until they demonstrate the requisite performance benchmark. Proficiency demonstration will be mandatory before progressing to ward proctored skill supervision on real patients. In addition, the doctors in training will receive ongoing and proximate feedback on their sampling mislabeling.
  Other Names: Medical Education; Simulation Training
  Arms: Control Group B; Interventional Group

SUMMARY:
The objective of this study is to determine the effectiveness of a Proficiency Based Progression training programme, together with evidence based individual feedback for any residual errors, which has been specifically developed for healthcare professionals performing phlebotomy at Cork University Hospital at reducing blood sampling errors including Wrong Blood in Tube (WBIT). This will allow us to internationally address the universal problem of sample mislabeling and WBIT. A pilot project which consisted of PBP delivered to 46 interns commencing work in July 2017 has shown a 47% reduction in haematology errors and a 67% reduction in WBITs in the haematology department. However, the sample size was small to result in a statistically significant reduction in WBITs and the investigators are concerned that the results were undermined by the fact that SHOs were not using the method outlined by the metric and may have influenced the standard practice of interns. This study by training interns and SHOs will be better able to determine the influence of the training programme in reducing error rates.

DETAILED DESCRIPTION:
Objective To determine the effectiveness of a Proficiency Based Progression Training programme, together with evidence based individual feedback for any residual errors, which has been specifically developed for healthcare professionals performing phlebotomy at Cork University Hospital at reducing blood sampling errors including Wrong Blood in Tube (WBIT) .The investigators will use the research data generated to recommend an evidence based training and competency assessment approach to health care providers in Ireland,. This will allow us to internationally address the universal problem of sample mislabeling and WBIT.

METHODS Subjects All SHO (128) and intern (46) trainees working at participating sites during an 18-month timeframe will be asked to participate. For interns the investigators will expect their participation in the two weeks before they commence work in June/July 2018/9. For SHO's the investigators will ensure training is integrated as part of their normal work routine and hospital practices. Participation will be expected and the investigators have secured the backing of the hospital executive management group, clinical directors and university teachers for implementation of this study.

Proficiency based progression training The phlebotomy metric which was developed at CUH in 2017 is the provides the key tool in the development of the PBP training programme. All interns and SHOs in institutions participating in the study will receive PBP training. All trainees will be required to engage with an online didactic education package and a simulation skill training module. Both of these education and training platforms will be derived from the procedure characterisation and benchmarked on experienced practitioner's performance. Trainees will be required to engage with the education and training platforms in a process of deliberate practice learning until they demonstrate the requisite performance benchmark. Only at that point will they be allowed to take samples in a clinical setting. Proficiency demonstration will be mandatory before progressing to ward proctored skill supervision on real patients. In addition, the doctors in training will receive ongoing and proximate feedback on their sampling mislabeling (including wrong blood in tube) performance as soon as it is discovered. Furthermore, they would be responsible for taking the new sample and explain to the patient the accurate reason why the blood sample had to be re-taken, as per open disclosure policy in the HSE.

Comparison Groups The control groups will be derived from extensive baseline data from CUH hospitals from trainees

Control group A: 1 -year historical data (2016/2017) The blood sampling error rate in the interns receiving PBP training in 2018 will be compared to historical data on doctors who would have received whatever training they would normally undergo as a part of their existing training program. It will not differ from what they would normally receive at that institution.

Control group B (2017/2018) In a pilot project in July 2017, 46 interns received the phlebotomy PBP training at CUH. The error rates in the interns in 2017 will be compared to the newly trained interns in 2018 to determine the effectiveness of the training over time.

Data collection at Cork University Hospital The Medically qualified clinical researcher Dr Noirin O'Herlihy, will set up and co-ordinate training for the two medical groups. She will inform the Interns and SHO in formal and informal sessions. She will be present at session to ensure accurate simulation of real life ward environments. She will obtain written informed consent from the medics in simulation and collect baseline demographic data on all doctors in training participating in the study.

Once competency has been demonstrated in simulation, she will be responsible for setting up real life clinical, monitored competency assessment in the real ward setting. Data collection will take place using an agreed standard operating procedure which is closely adhered to by all data collection sites.

ELIGIBILITY:
Inclusion Criteria:

All blood samples performed at Cork Unversity Hospital and Kerry General Hospital by Doctors in Training

Exclusion Criteria:

If the doctor is not using his own log in to request blood samples on the clinical manager software If the doctor does not attend the training session

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Total Number of Rejected Samples due to pre-analytical errors | 6 months
  The total number of blood samples that were not tested due to pre analytical errors by the doctors in training as a percentage of the total number of samples taken by the doctors

SECONDARY OUTCOMES:
Over and Underfilling of the specimen bottle | 6 months
  Any sample not tested due to over or under filling of the bottle as a percentage of the total number of samples performed
Clotted Samples | 6 months
  The number of samples not tested due to clotting of the sampleas a percentage of the total number of samples performed
Haemolysed Samples | 6 months
  The number of blood samples not tested as the blood sample was haemolysedas a percentage of the total number of samples performed
No Specimen Received | 6 months
  The number of blood requests received without a specimen bottleas a percentage of the total number of samples performed
Incorrect Bottle | 6 months
  The number of blood requests received where the blood was taken in the incorrect specimen bottle as a percentage of the total number of samples performed
Other Causes for Rejected Samples | 6 months
  Any other cause for the blood request not being processed as a percentage of the total number of samples performed
Wrong Blood in Tube | 6 months
  The number of specimens where the blood sample in the tube is not that of the patient label on the specimen bottle as a percentage of the total number of samples performed

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Gallagher, PhD, Study Director — University College Cork; Mary R Cahill, MD, Principal Investigator — University College Cork
Locations (1):
- Cork University Hospital, Cork, Munster, Ireland

IPD SHARING:
Plan to Share IPD: Yes
The study data will be made available once the study is completed by contacting the principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18 months
Access Criteria: At completion of the study